CLINICAL TRIAL: NCT05674721
Title: A Randomized, Open Label, Single Center, Single Dose, Two Treatment, Two Period, Two Sequence Crossover Bioequivalence Study of Advil PM Liqui-Gels Minis (Ibuprofen/Diphenhydramine Hydrochloride 200 mg/25 mg) To Advil PM Liqui-Gels (Ibuprofen/Diphenhydramine Hydrochloride 200 mg/25 mg) in Healthy Adult Subjects Under Fasted Conditions
Brief Title: A Bioequivalence Study of Advil PM Liqui-Gels Minis (Ibuprofen/Diphenhydramine Hydrochloride 200 mg/25 mg) Compared to the Current Marketed Advil PM Liqui-Gels (Ibuprofen/Diphenhydramine Hydrochloride 200 mg/25 mg) in Healthy Adult Subjects Under Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 218677
Record Dates: First submitted 2022-12-16; First posted 2023-01-06 (Actual); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advil PM Liqui-Gels Minis (Experimental): Participants will be randomly assigned as per cross-over design to receive a single dose of 2 Advil PM Liqui-Gels Minis capsules orally on day 1 of period 1 and will receive single dose of 2 Advil PM Liqui-Gels capsules orally on day 1 of period 2 with at least 7 days washout period. Participants will be instructed to consume the entire amount of ambient temperature water (approximately 240 milliliters [mL]) along their investigational product.
  Interventions: Drug: Advil PM Liqui-Gels Minis
- Advil PM Liqui-Gels (Active Comparator): Participants will be randomly assigned as per cross-over design to receive a single dose of 2 Advil PM Liqui-Gels capsules orally on day 1 of period 1 and will receive single dose of 2 Advil PM Liqui-Gels Minis capsules orally on day 1 of period 2 with at least 7 days washout period. Participants will be instructed to consume the entire amount of ambient temperature water (approximately 240 mL) along their investigational product.
  Interventions: Drug: Advil PM Liqui-Gels

INTERVENTIONS:
Drug: Advil PM Liqui-Gels Minis — Ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg, Oral capsule which is a size reduction of the currently marketed reference product.
  Arms: Advil PM Liqui-Gels Minis
Drug: Advil PM Liqui-Gels — Ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg, Oral capsule.
  Arms: Advil PM Liqui-Gels

SUMMARY:
The purpose of this study is to support the submission of Advil PM Liqui-Gels Minis (ibuprofen/diphenhydramine hydrochloride 200 milligrams [mg]/25 mg) which is a size reduction of the currently marketed Advil PM Liqui-Gels, by determining if this product is bioequivalent to the reference product Advil PM Liqui-Gels (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg) under fasting conditions.

DETAILED DESCRIPTION:
This is a single center, single dose, open-label, randomized, two-treatment, two-sequence, two-period crossover, bioequivalence study in healthy adult participants with at least a 7-day washout period. A sufficient number of participants will be screened to randomize approximately 44 to ensure at least 37 evaluable participants complete the entire study. Participants will be randomly assigned to one of 2 treatment sequences and receive a single dose of one of the treatments in each period following a crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Participant who is willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Healthy participant, which is defined as in general good physical health, as judged by the investigator and no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead Electrocardiogram (ECG) or clinical laboratory tests.
* Body Mass Index (BMI) of 18.5 to 30.0 Kilogram per meter square (kg/m^2); and a total body weight greater than or equal to (>=)50.0 Kilogram (kg) for males and >=45.0 kg for females.
* Female participant of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study and for at least 30 days after the last dose of assigned treatment. Female participant who is not of childbearing potential must meet at least one of the following criteria: A. Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle-stimulating hormone (FSH) level >= 40 mili international unit per milliliter (mIU/mL) B. Have undergone a documented (including self-reported) hysterectomy and/or bilateral oophorectomy.
* Participant with two negative tests (one at screening within 72 hours of admission and one at check in Day-1 in Period 1) for active coronavirus disease 2019 (COVID-19), separated by more than (>)24 hours.

Exclusion Criteria:

* Participant who is an investigational site staff member directly involved in the conduct of the study and his/her family members, site staff member otherwise supervised by the Investigator, or participant who is a GlaxoSmithKline (GSK) employee directly involved in the conduct of the study.
* Participation in other studies involving investigational drug(s) within 30 days prior to study entry and/or during study participation.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Pregnant female participant as confirmed by a positive pregnancy test or intending to become pregnant over the duration of the study.
* Breastfeeding female participant.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients (gelatin, medium-chain triglycerides, pharmaceutical ink, polyethylene glycol, potassium hydroxide, purified water, sorbitol sorbitan solution).
* Any history of asthma, urticaria, or other significant allergic diathesis or allergic reaction to any other pain reliever/fever reducer. Participant with uncomplicated seasonal allergic rhinitis can be accepted if expected allergy season is clearly outside enrollment/treatment period.
* Diagnosis of long QT syndrome or QTcF > 450 millisecond (msec) for males and > 470 msec for females at screening.
* Clinically significant vital sign abnormalities (systolic blood pressure lower than 90 or over 140 millimeters of mercury [mmHg], diastolic blood pressure lower than 50 or over 90 mmHg, or pulse rate less than 50 or over 100 beats per minute [bpm]).
* Unwilling or unable to comply with the Lifestyle Considerations described in this protocol.
* Use of any medication (including over the counter [OTC] medications and herbal remedies) within 2 weeks or within less than 10 times the elimination half-life of the respective drug (whichever is longer) before first scheduled study drug administration or is anticipated to require any concomitant medication during that period or at any time throughout the study. Allowed treatments are:

  1. systemic contraceptives and hormone replacement therapy, as long as female participant is on stable treatment for at least 3 months before first scheduled study drug administration and continues treatment throughout the study.
  2. occasional use of acetaminophen (up to 2 grams [g] daily).
* Evidence or history of clinically significant laboratory abnormality, hematological, renal, endocrine, pulmonary, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease within the last 5 years that may increase the risk associated with study participation.
* Clinically relevant chronic or acute infectious illnesses or febrile infections within two weeks prior to start of the study.
* Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance but not limited to any of the following:

  1. History of major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, bowel resection, gastric bypass, gastric stapling or gastric banding (note: this is not applicable for minor abdominal surgery without significant tissue resection, for example, appendectomy and herniorrhaphy).
  2. History of inflammatory bowel disease or gastrointestinal bleeding including peptic ulcers.
  3. History or current evidence of renal disease or impaired renal function at screening as indicated by abnormal levels of serum creatinine (> 1.43 milligram/deciliter [mg/dL]) or blood urea nitrogen (BUN) (>= 35 mg/dL) or the presence of clinically significant abnormal urinary constituents (e.g., albuminuria).
  4. History or current evidence of ongoing hepatic disease or impaired hepatic function at screening. A participant will be excluded if more than one of the following lab value deviations are found: 1) Aspartate aminotransferase (AST) (>= 1.2 upper limit of normal [ULN]), Alanine transaminase (ALT) (>= 1.2 ULN), 2) Gamma-glutamyl transferase (GGT) (>= 1.2 ULN), Alkaline phosphatase (ALP) (>= 1.2 ULN), 3) total bilirubin (> 2.00 mg/dL) or creatine kinase (>= 3 ULN). A single deviation from the above values is acceptable and will not exclude the candidate, unless specifically advised by the investigator.
  5. Evidence of urinary obstruction (for example, due to benign prostate hyperplasia) or difficulty in voiding at screening.
  6. Diagnosis of angle-closure (narrow angle) glaucoma.
  7. History or clinical evidence at screening of pancreatic injury or pancreatitis.
* Participant with signs and symptoms suggestive of COVID-19 (for example, fever, cough, and so on within 14 days of inpatient admission as defined by World Health Organization (WHO) or local guidance.
* Participant with known COVID-19 positive contacts in the past 14 days.
* Any vaccination, including COVID-19 vaccine, within 14 days prior to the first dose.
* History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
* History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5 percent [%], 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* Positive urine drug screen or alcohol breath test at screening.
* Participant reported regular consumption of beverages or food containing xanthine derivatives or xanthine-related compounds (for example, coffee, tea, caffeine-containing sodas and chocolate), equivalent to >= 500 mg xanthine per day.
* Current smoker, defined as the use of tobacco or nicotine products during the 3 months prior to screening until admission to the unit or a positive urine cotinine test at screening.
* Participant reports consumption of any drug metabolizing enzyme (e.g., CYP3A4 or other cytochrome P450 enzymes) inducing or inhibiting aliments, beverages or food supplements (for example, broccoli, Brussels sprouts, grapefruit, grapefruit juice, star fruit, St. John's Wort and so on) within 2 weeks prior to admission to the unit.
* Performance of strenuous physical exercise (body building, high performance sports) from 2 weeks prior to admission and throughout the entire study.
* Allergy to skin disinfecting agents, tape, or latex rubber, whenever appropriate substitutions cannot be applied or in the Investigator's opinion may pose a risk to the Participant.
* Any condition not identified in the protocol that in the opinion of the investigator would confound the evaluation and interpretation of the study data or may put the participant at risk.
* Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to dosing.
* Hemoglobin value less than (<)12.0 grams per deciliter (g/dL) for males and < 11.5 g/dL for females.
* Participant who has previously been enrolled in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2023-01-05 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data and study documents can be requested for further research from ww.clinical-trial-register@haleon.com
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at a single center in the United States.
Pre-assignment Details: A total of 144 participants were screened of which 77 were enrolled. Of the 77 enrolled participants, 33 were not randomized and 44 were randomized as per cross-over design to one of the two treatment sequences: Sequence AB (Advil PM Liqui-Gels Minis followed by Advil PM Liqui-Gels) or Sequence BA (Advil PM Liqui-Gels followed by Advil PM Liqui-Gels Minis). A total of 42 participants completed the study.
Groups:
- Sequence AB: Advil PM Liqui-Gels Minis Followed by Advil PM Liqui-Gels: Participants received a single dose of 2 Advil PM Liqui-Gels Minis (ibuprofen/diphenhydramine hydrochloride 200 milligrams [mg]/25 mg), capsules, orally on Day 1 of Treatment Period 1 under fasted conditions as Treatment A followed by a single dose of 2 Advil PM Liqui-Gels (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Period 2 under fasted conditions as Treatment B. There was a washout period of at least 7 days between each dosing. Participants were instructed to consume the entire amount of ambient temperature water (approximately 240 milliliters [mL]) along with their investigational product.
- Sequence BA: Advil PM Liqui-Gels Followed by Advil PM Liqui-Gels Minis: Participants received a single dose of 2 Advil PM Liqui-Gels (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Period 1 under fasted conditions as Treatment B followed by a single dose of 2 Advil PM Liqui-Gels Minis (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Period 2 under fasted conditions as Treatment A. There was a washout period of at least 7 days between each dosing. Participants were instructed to consume the entire amount of ambient temperature water (approximately 240 mL) along with their investigational product.
Period: Treatment Period 1 (Up to 3 Days)
Arm/Group | Sequence AB: Advil PM Liqui-Gels Minis Followed by Advil PM Liqui-Gels | Sequence BA: Advil PM Liqui-Gels Followed by Advil PM Liqui-Gels Minis
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Washout Period (Up to 7 Days)
Arm/Group | Sequence AB: Advil PM Liqui-Gels Minis Followed by Advil PM Liqui-Gels | Sequence BA: Advil PM Liqui-Gels Followed by Advil PM Liqui-Gels Minis
Started | 22 | 22
Completed | 22 | 20
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Treatment Period 2 (Up to 3 Days)
Arm/Group | Sequence AB: Advil PM Liqui-Gels Minis Followed by Advil PM Liqui-Gels | Sequence BA: Advil PM Liqui-Gels Followed by Advil PM Liqui-Gels Minis
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was defined as all randomized participants who received at least one dose of study medication.
Groups:
- Sequence AB: Advil PM Liqui-Gels Minis Followed by Advil PM Liqui-Gels: Participants received a single dose of 2 Advil PM Liqui-Gels Minis (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Period 1 under fasted conditions as Treatment A followed by a single dose of 2 Advil PM Liqui-Gels (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Period 2 under fasted conditions as Treatment B. There was a washout period of at least 7 days between each dosing. Participants were instructed to consume the entire amount of ambient temperature water (approximately 240 mL) along with their investigational product.
- Total: Total of all reporting groups
Arm/Group | Sequence AB: Advil PM Liqui-Gels Minis Followed by Advil PM Liqui-Gels | Sequence BA: Advil PM Liqui-Gels Followed by Advil PM Liqui-Gels Minis | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (7.02) | 33.7 (9.76) | 33.4 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 22 | 44
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 5 | 4 | 9
  White | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Ibuprofen
Description: Cmax was defined as maximum observed post-dose plasma concentration for ibuprofen obtained without interpolation. Blood samples were collected at indicated timepoints and pharmacokinetic (PK) analysis was performed. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported.
Time Frame: 1 hour prior to dosing (pre-dose) and at 10,15,30,45 minutes and 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5, 6, 8,10,12 and 16 hours post-dose on Day 1 (First Intervention) and Day 11 (Second Intervention)
Population: PK analysis set included all participants of the PK population who completed both Treatment Periods, and for which the relevant PK parameters (at least one area under the curve [AUC] or Cmax) could be derived. The PK population was defined as all randomized participants who had at least one post-dose PK value, and who had no major protocol deviations concerning PKs.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A (Test): Participants received a single dose of 2 Advil PM Liqui-Gels Minis (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Periods 1 and 2 under fasted conditions as Treatment A.
- Treatment B (Reference): Participants received a single dose of 2 Advil PM Liqui-Gels (ibuprofen/diphenhydramine hydrochloride 200 mg/25 mg), capsules, orally on Day 1 of Treatment Periods 1 and 2 under fasted conditions as Treatment B.
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
nanogram per milliliter (ng/mL) | 36879.50 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 25.2 | 38875.03 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 18.0
Statistical Analysis 1: Comparison: Treatment A (Test) vs Treatment B (Reference); Test type: Equivalence — The bioequivalence between Treatment A (test) and Treatment B (reference) under fasted conditions would be declared as per Food and Drug Administration (FDA) requirements if the 90 percent (%) confidence intervals (CIs) for the ratio of the geometric means of Cmax were between 80% and 125%; Ratio of Geometric Least Square Mean = 95.13, 90% CI 2-sided [88.31 to 102.47]

2. Primary Outcome: Cmax for Diphenhydramine
Description: Cmax was defined as maximum observed post-dose plasma concentration for diphenhydramine obtained without interpolation. Blood samples were collected at indicated timepoints and PK analysis was performed. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported.
Time Frame: 1 hour prior to dosing (pre-dose) and at 10,15,30,45 minutes and 1,1.25,1.5,1.75,2,2.25,2.5,2.75,3, 3.25, 3.5, 3.75, 4, 4.25, 4.5, 4.75, 5, 5.25, 5.5,6,8,10,12,16,24,36, and 48 hours post-dose on Day 1 (First Intervention) and Day 11 (Second Intervention)
Population: PK analysis set. Here, overall number analyzed is defined as the number of participants with data available for analysis for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
ng/mL | 75.40 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 40.5 | 73.22 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 40.0
Statistical Analysis 1: Comparison: Treatment A (Test) vs Treatment B (Reference); Test type: Equivalence — The bioequivalence between Treatment A (test) and Treatment B (reference) under fasted conditions would be declared as per FDA if the 90% CIs for the ratio of the geometric means of Cmax were between 80% and 125%; Ratio of Geometric Least Square Mean = 102.51, 90% CI 2-sided [93.54 to 112.35]

3. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated From Time 0 to the Last Measurable Sampling Time Point (t) (AUC [0-t]) for Ibuprofen
Description: AUC (0-t) was defined as the area under the plasma concentration versus time curve calculated from time zero to the last measurable sampling time point, (t) using linear up log down trapezoidal method. Blood samples were collected at indicated timepoints and PK analysis was performed. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per milliliter (h*ng/ mL)
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
hour*nanogram per milliliter (h*ng/ mL) | 121612.36 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 22.3 | 123012.43 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 20.7
Statistical Analysis 1: Comparison: Treatment A (Test) vs Treatment B (Reference); Test type: Equivalence — The bioequivalence between Treatment A (test) and Treatment B (reference) under fasted conditions would be declared as per FDA if the 90% CIs for the ratio of the geometric means of AUC0-t were between 80% and 125%; Ratio of Geometric Least Square Mean = 99.15, 90% CI 2-sided [96.76 to 101.61]

4. Primary Outcome: AUC (0-t) for Diphenhydramine
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
h*ng/mL | 746.76 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 49.2 | 728.13 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 49.7
Statistical Analysis 1: Comparison: Treatment A (Test) vs Treatment B (Reference); Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of Geometric Least Square Mean = 102.62, 90% CI 2-sided [98.15 to 107.30]

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve Calculated From Time 0 to Infinity (AUC [0-inf]) for Ibuprofen
Description: AUC (0-inf) was defined as area under the plasma concentration versus time curve calculated from time 0 to infinity, computed as AUC0-inf = AUC0-t + C(last)/λz where C(last) was the concentration at the last measurable sampling time point and λz was the terminal elimination rate constant. Blood samples were collected at indicated timepoints and PK analysis was performed. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
h*ng/mL | 123067.92 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 22.2 | 124401.36 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 20.7
Statistical Analysis 1: Comparison: Treatment A (Test) vs Treatment B (Reference); Test type: Equivalence — The bioequivalence between Treatment A (test) and Treatment B (reference) under fasted conditions would be declared as per FDA if the 90% CIs for the ratio of the geometric means of AUC0-inf were between 80% and 125%; Ratio of Geometric Least Square Mean = 99.20, 90% CI 2-sided [96.82 to 101.63]

6. Primary Outcome: AUC (0-inf) for Diphenhydramine
Description: AUC (0-inf) was defined as area under the plasma concentration versus time curve calculated from time 0 to infinity computed as AUC0-inf = AUC0-t + C(last)/λz where C(last) was the concentration at the last measurable sampling time point and λz was the terminal elimination rate constant. Blood samples were collected at indicated timepoints and PK analysis was performed. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
h*ng/mL | 782.89 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 52.3 | 762.79 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (CV%) is being reported. CV% = 52.7
Statistical Analysis 1: Comparison: Treatment A (Test) vs Treatment B (Reference); Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Ratio of Geometric Least Square Mean = 102.73, 90% CI 2-sided [98.31 to 107.34]

7. Secondary Outcome: Terminal Elimination Rate Constant (λz) for Ibuprofen
Description: λz was computed as negative of the estimated slope of the linear regression of the ln-transformed concentration versus time profile in the terminal elimination phase. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
1/hour | 0.3252 (0.05931) | 0.3329 (0.06812)

8. Secondary Outcome: λz for Diphenhydramine
Description: λz was computed as the negative of the estimated slope of the linear regression of the ln-transformed concentration versus time profile in the terminal elimination phase. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
1/hour | 0.0665 (0.01342) | 0.0669 (0.01277)

9. Secondary Outcome: Time of the Maximum Observed Post-dose Concentration (Tmax) for Ibuprofen
Description: tmax was defined as time of the maximum observed post-dose concentration. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
hour | 1.000 [0.250 to 4.750] | 0.875 [0.500 to 3.250]

10. Secondary Outcome: Tmax for Diphenhydramine
Description: as for outcome 9
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
hour | 3.000 [1.500 to 5.500] | 3.000 [2.000 to 5.000]

11. Secondary Outcome: The Elimination Half-life (t1/2) for Ibuprofen
Description: Elimination half-life was computed as t1/2 = ln(2)/λz where λz is the terminal elimination rate constant. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
hour | 2.21 [1.34 to 3.07] | 2.04 [1.49 to 4.40]

12. Secondary Outcome: t1/2 for Diphenhydramine
Description: as for outcome 11
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
hour | 10.71 [6.29 to 14.41] | 10.45 [6.39 to 14.85]

13. Secondary Outcome: Apparent Volume of Distribution (Vz/F) for Ibuprofen
Description: Vz/F was calculated by the dose administered/(λz*AUC0-inf) where λz was the terminal elimination rate constant and AUC0-inf was area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
liter | 10.35 (2.06) | 10.17 (2.56)

14. Secondary Outcome: Vz/F for Diphenhydramine
Description: Vz/F was calculated by the dose administered/(λz*AUC0-inf) where λz is the terminal elimination rate constant and AUC0-inf is area under the plasma concentration versus time curve calculated from time 0 to infinity. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
liter | 1059.73 (449.56) | 1071.75 (411.77)

15. Secondary Outcome: Apparent Total Clearance (CI/F) for Ibuprofen
Description: CI/F was calculated as dose administered/AUC0-inf where AUC0-inf was area under the plasma concentration versus time curve calculated from time zero to infinity. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 1
Population: PK analysis set.
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 42
liter per hour | 3.33 (0.75) | 3.28 (0.65)

16. Secondary Outcome: CI/F for Diphenhydramine
Description: CI/F was calculated as dose administered/ AUC0-inf where AUC0-inf was area under the plasma concentration versus time curve calculated from time zero to infinity. Blood samples were collected at indicated timepoints and PK analysis was performed.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter per hour
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 41 | 41
liter per hour | 71.95 (37.05) | 72.85 (33.18)

17. Secondary Outcome: Number of Participants Reporting Ease of Swallowing on 5-Point Ordinal Scale
Description: Immediately after dosing, the assessment of 'ease of swallowing' was done via one question with an ordinal response (ease of swallowing on 5-point ordinal scale) of each product. Participants ranked the 'ease of swallowing' of the product on a scale from 1 to 5 where 1=not easy to swallow; 2=somewhat easy to swallow; 3=average to swallow; 4=above average to swallow; 5=very easy to swallow. Higher score indicated more ease in swallowing.
Time Frame: Post-dose on Day 1 (First Intervention) and Day 11 (Second Intervention)
Population: The safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A (Test) | Treatment B (Reference)
Number analyzed (Participants) | 42 | 44
Participants
  1 (Not Easy to Swallow) | 0 | 0
  2 (Somewhat Easy to Swallow) | 0 | 0
  3 (Average to Swallow) | 0 | 1
  4 (Above Average to Swallow) | 1 | 3
  5 (Very Easy to Swallow) | 41 | 40

ADVERSE EVENTS:
Time Frame: From screening up to end of study (up to 38 days)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device). A Serious Adverse Event (SAE) is a particular category of an adverse event where the adverse outcome is serious.
Arm/Group | Treatment A (Test) | Treatment B (Reference)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/44
Other Adverse Events (participants affected / at risk) | 3/42 | 5/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (Test) (N=42) | Treatment B (Reference) (N=44)
Haemoglobin decreased (Investigations) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 2
Catheter site pain (General disorders) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT05674721/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT05674721/SAP_001.pdf